CLINICAL TRIAL: NCT01618162
Title: The Efficacy of Insulin Degludec/Liraglutide as add-on Therapy in Controlling Glycaemia in Adults With Type 2 Diabetes Inadequately Controlled on Sulphonylurea With or Without Metformin Therapy
Acronym: DUAL™IV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9068-3951; 2012-000140-97 (EudraCT Number); U1111-1126-9776 (Other: WHO)
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin degludec/liraglutide (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Injected subcutaneously (under the skin) once daily. Dose individually adjusted.
  Arms: Insulin degludec/liraglutide
Drug: placebo — Injected subcutaneously (under the skin) once daily.
  Arms: Placebo

SUMMARY:
This trial is conducted in Asia, Europe and the United States of America (USA). The aim of this trial is to investigate the efficacy and safety of insulin degludec/liraglutide in insulin naïve subjects inadequately controlled with SU (sulphonylurea) alone or in combination with metformin. All subjects will continue their pre-trial SU treatment with or without metformin treatment without changing the frequency or dose throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus
* HbA1c 7.0-9.0% (53-75 mmol/mol) (both inclusive)
* Subjects on stable daily dose of sulphonylurea (above or equal to half of the max approved dose according to local label) with or without metformin (above or equal to 1500 mg or max tolerated dose) for at least 90 days prior to screening visit (Visit 1)
* Body Mass Index (BMI) below or equal to 40 kg/m^2

Exclusion Criteria:

* Any use of oral anti-diabetic drugs (OADs) (other than SU in monotherapy or in combinationwith metformin) below or equal to 90 days prior to screening visit (Visit 1)
* Use of any drug (other than SU in monotherapy or in combination with metformin), which in the Investigators opinion could interfere with the blood glucose level (e.g. systemic corticosteroids)
* Previous treatment with glucagon-like peptide-1 (GLP-1) receptor agonist (e.g. exenatide, liraglutide)
* Treatment with any insulin regimen (short term treatment due to intercurrent illness including gestational diabetes is allowed at the discretion of the Investigator)
* Screening calcitonin above or equal to 50 ng/l
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2)
* Cardiovascular disorders defined as: congestive heart failure (New York Heart Association (NYHA) class III-IV), diagnosis of unstable angina pectoris, cerebral stroke and/or myocardial infarction within the past 52 weeks prior to screening visit (Visit 1) and/or planned coronary,carotid or peripheral artery revascularisation procedures
* Proliferative retinopathy requiring acute treatment or maculopathy (macular oedema) according to the Investigator's opinion
* Subjects with a clinical significant, active (during the past 12 months) disease of the gastrointestinal, pulmonary, endocrinological (except for the Type 2 Diabetes Mellitus),neurological, genitourinary or haematological system that in the opinion of the Investigator,may confound the results of the trial or pose additional risk in administering trial product
* History of chronic pancreatitis or idiopathic acute pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2012-08-29 (Actual); Primary Completion 2013-10-23 (Actual); Study Completion 2013-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (82):
- United States (42):
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Garden Grove, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Crestview Hills, Kentucky
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Saint Charles, Missouri
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Lodi, New Jersey
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Tabor City, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Pelzer, South Carolina
  - Novo Nordisk Investigational Site, Simpsonville, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
- Bulgaria (3):
  - Novo Nordisk Investigational Site, Lukovit
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sofia
- Canada (10):
  - Novo Nordisk Investigational Site, Burnaby, British Columbia
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Victoria, British Columbia
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Mirabel, Quebec
  - Novo Nordisk Investigational Site, Pointe-Claire, Quebec
  - Novo Nordisk Investigational Site, Sherbrooke, Quebec
  - Novo Nordisk Investigational Site, Québec
- Germany (7):
  - Novo Nordisk Investigational Site, Esslingen am Neckar
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Sulzbach-Rosenberg
- India (7):
  - Novo Nordisk Investigational Site, Guwahati, Assam
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Belagavi, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Delhi, New Delhi
  - Novo Nordisk Investigational Site, Hyderabad
- Israel (7):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Novo Nordisk Investigational Site, Manatí, Puerto Rico
- Turkey (Türkiye) (5):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Gaziantep
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir

REFERENCES:
- [Background] Khunti K, Mohan V, Jain SM, Boesgaard TW, Begtrup K, Sethi B. Efficacy and Safety of IDegLira in Participants with Type 2 Diabetes in India Uncontrolled on Oral Antidiabetic Drugs and Basal Insulin: Data from the DUAL Clinical Trial Program. Diabetes Ther. 2017 Jun;8(3):673-682. doi: 10.1007/s13300-017-0252-9. Epub 2017 Mar 22. PMID 28332144
- [Result] Rodbard HW, Bode BW, Harris SB, Rose L, Lehmann L, Jarlov H, Thurman J; Dual Action of Liraglutide and insulin degludec (DUAL) IV trial investigators. Safety and efficacy of insulin degludec/liraglutide (IDegLira) added to sulphonylurea alone or to sulphonylurea and metformin in insulin-naive people with Type 2 diabetes: the DUAL IV trial. Diabet Med. 2017 Feb;34(2):189-196. doi: 10.1111/dme.13256. Epub 2016 Oct 7. PMID 27589252
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 77 sites in 7 countries: Bulgaria (7), Canada (9), Germany (6), India (6), Israel (7), Turkey (3), United States (39).
Pre-assignment Details: The trial included a 2 week screening period to assess subject eligibility.
Groups:
- IDegLira: In this arm, subjects suboptimally controlled on sulfonyl urea (SU) +/- metformin, were given subcutenaous (s.c.) injection of insulin degludec/liraglutide (IDegLira). SU and metformin were maintained at the stable pre-trial dose throughout the duration of the trial. IDegLira was injected in the thigh, upper arm (deltoid region) or abdomen once daily preferably at the same time every day. The injection area chosen remained unchanged throughout the trial, but rotation within the area was recommended. Treatment with IDegLira was initiated at 10 dose steps containing 10 units insulin degludec and 0.36 mg liraglutide. Adjustment of the IDegLira dose was performed twice weekly based on the mean of 3 preceding daily fasting SMPG values on 3 consecutive days (fasting glycaemic target of 4.0-6.0 mmol/L).
- Placebo: In this arm, subjects suboptimally controlled on SU +/- metformin, were given s.c. injection of placebo solution (matched to IDegLira) and was initiated and titrated as described for IDegLira. SU and metformin were maintained at the stable pre-trial dose throughout the duration of the trial. Placebo solution was injected in the thigh, upper arm (deltoid region) or abdomen once daily preferably at the same time every day. The injection area chosen remained unchanged throughout the trial, but rotation within the area was recommended. Adjustment of placebo was performed twice weekly based on the mean of 3 preceding daily fasting SMPG values on 3 consecutive days (fasting glycaemic target of 4.0-6.0 mmol/L).
Period: Overall Study
Arm/Group | IDegLira | Placebo
Started | 289 | 146
Exposed | 288 | 146
Completed | 251 | 111
Not Completed | 38 | 35
Not completed — Protocol Violation | 13 | 10
Not completed — Adverse Event | 9 | 2
Not completed — Withdrawal Criteria | 2 | 10
Not completed — Unclassified | 14 | 13

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized subjects.
Groups:
- IDegLira: In this arm, Subjects suboptimally controlled on SU +/- metformin, were given s.c. injection of IDegLira. SU and metformin were maintained at the stable pre-trial dose throughout the duration of the trial. IDegLira was injected in the thigh, upper arm (deltoid region) or abdomen once daily preferably at the same time every day. The injection area chosen remained unchanged throughout the trial, but rotation within the area was recommended. Treatment with IDegLira was initiated at 10 dose steps containing 10 units insulin degludec and 0.36 mg liraglutide. Adjustment of the IDegLira dose was performed twice weekly based on the mean of 3 preceding daily fasting SMPG values on 3 consecutive days (fasting glycaemic target of 4.0-6.0 mmol/L).
- Total: Total of all reporting groups
Arm/Group | IDegLira | Placebo | Total
Number analyzed (Participants) | 289 | 146 | 435
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.6) | 59.4 (10.8) | 59.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 73 | 208
  Male | 154 | 73 | 227
Glycosylated haemoglobin [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.9 (0.6) | 7.9 (0.6) | 7.9 (0.6)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] | 9.1 (2.2) | 9.1 (2.1) | 9.1 (2.1)
Body weight [Mean (Standard Deviation); unit: kilograms] | 87.2 (18.6) | 89.3 (17.5) | 87.9 (18.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline to 26 weeks.
Time Frame: Week 0, Week 26
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegLira | Placebo
Number analyzed (Participants) | 289 | 146
percentage of glycosylated haemoglobin | -1.45 (0.84) | -0.46 (0.83)
Statistical Analysis 1: Comparison: IDegLira vs Placebo; Superiority of IDegLira versus placebo therapy would be concluded if the 95% CI for the treatment differences for change in HbA1c lied entirely below 0%; implying that the two-sided p-value calculated by the ANCOVA model for testing the hypothesis of no difference between treatments was less than 5%; Test type: Superiority or Other; p < 0.001, ANCOVA; Estimated treatment difference = -1.02, 95% CI 2-sided [-1.18 to -0.87]

2. Secondary Outcome: Responders Achieving Pre-defined Target: HbA1c Below 7.0% (53 mmol/Mol)
Description: Percentage of subjects having HbA1c below 7% at week 26.
Time Frame: Week 26
Population: Full analysis set.
Measure: Number; unit: percentage of subjects
Arm/Group | IDegLira | Placebo
Number analyzed (Participants) | 289 | 146
percentage of subjects | 79.2 | 28.8

3. Secondary Outcome: Responders Achieving Pre-defined Target: HbA1c Below or Equal to 6.5% (48 mmol/Mol)
Description: Percentage of subjects having HbA1c below 6.5% at week 26
Time Frame: Week 26
Population: Full analysis set.
Measure: Number; unit: percentage of subjects
Arm/Group | IDegLira | Placebo
Number analyzed (Participants) | 289 | 146
percentage of subjects | 64 | 12.3

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG at week 26.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of subjects analyzed=subjects with data available for FPG.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegLira | Placebo
Number analyzed (Participants) | 286 | 144
mmol/L | -2.6 (2.61) | -0.31 (2.43)

5. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight at week 26.
Time Frame: Week 0, week 26
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | IDegLira | Placebo
Number analyzed (Participants) | 289 | 146
kilogram | 0.5 (3.1) | -1 (2.6)

6. Secondary Outcome: Number of Treatment Emergent (Confirmed) Hypoglycaemic Episodes
Description: An event was treatment emergent if the onset of the episode occurs after the first administration of trial product and no later than 7 days after last trial product administration.
  Confirmed hypoglycaemic episodes were defined as hypoglycaemic episodes that were either severe or minor.
  Minor hypoglycaemic episodes were defined as:
  1. An episode with symptoms consistent with hypoglycaemia and confirmed by blood glucose value <2.8 mmol/L (50 mg/dL) or plasma glucose <3.1 mmol/L (56 mg/dL) and which was handled by the subject himself/herself.
  2. Any asymptomatic PG value <3.1 mmol/L (56 mg/dL) or blood glucose value <2.8 mmol/L (50 mg/dL).
  Severe hypoglycemia was defined as an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
  Reported values are hypoglycemia event rate per 100 patient-years of exposure (PYE).
Time Frame: After 26 weeks of treatment
Population: Safety analysis set included all subjects receiving at least one dose of the trial product.
Measure: Number; unit: event rate per 100 PYE
Arm/Group | IDegLira | Placebo
Number analyzed (Participants) | 288 | 146
event rate per 100 PYE | 351.7 | 135.2

7. Secondary Outcome: Number of Adverse Events (AEs)
Description: An AE was any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. Reported values are hypoglycemia event rate per 100 PYE.
Time Frame: After 26 weeks of treatment
Population: Safety analysis set.
Measure: Number; unit: event rate per 100 PYE
Arm/Group | IDegLira | Placebo
Number analyzed (Participants) | 288 | 146
event rate per 100 PYE | 401.4 | 367

ADVERSE EVENTS:
Time Frame: After 26 weeks of treatment
Description: Safety analysis set included 434 subjects (288 in IDegLira and 146 in placebo).
Arm/Group | IDegLira | Placebo
Serious Adverse Events (participants affected / at risk) | 14/288 | 5/146
Other Adverse Events (participants affected / at risk) | 83/288 | 38/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=288) | Placebo (N=146)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Meningitis haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Normal tension glaucoma (Eye disorders) | 1 (1) | 0 (0)
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=288) | Placebo (N=146)
Dyslipidaemia (Metabolism and nutrition disorders) | 19 (19) | 6 (7)
Headache (Nervous system disorders) | 15 (18) | 8 (11)
Influenza (Infections and infestations) | 8 (8) | 8 (9)
Lipase increased (Investigations) | 27 (29) | 6 (8)
Nasopharyngitis (Infections and infestations) | 25 (29) | 12 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone pubication and/or communication for up to 60 days to protect intellectual property.